CLINICAL TRIAL: NCT03753750
Title: Evaluation of Noninvasive Spinal Cord Stimulation for Neurogenic and Idiopathic Overactive Bladder
Brief Title: Noninvasive Spinal Cord Stimulation for Neurogenic and Idiopathic Overactive Bladder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment due to COVID-19 pandemic
Sponsor: University of Southern California (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Evgeniy I. Kreydin, Assistant Professor of Urology, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-18-00382
Record Dates: First submitted 2018-11-19; First posted 2018-11-27 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Overactive Bladder; Incontinence, Urge; Neurogenic Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge; Urinary Bladder, Neurogenic

STUDY DESIGN:
Intervention Model Description: Blinded sham-controlled trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Actual stimulation (Experimental): Subjects enrolled in the
  Interventions: Device: Noninvasive spinal cord stimulation
- Sham stimulation (Sham Comparator)
  Interventions: Device: Noninvasive spinal cord stimulation

INTERVENTIONS:
Device: Noninvasive spinal cord stimulation — Noninvasive spinal cord stimulation is a transcutaneous technique used to modulate the activity of the spinal cord. Subjects will undergo sham or actual stimulation 3-4 times a week for one hour at a time.

SUMMARY:
Overactive bladder (OAB) affects 12-30% of the world's population. The accompanying urinary urgency, urinary frequency and incontinence can impair the ability to work, interact in social activities and can result in poor social functioning. Multiple treatment modalities are available for overactive bladder. However, each therapy has drawbacks that limit its application in certain patient populations. For example, oral medications have significant side effects and suffer from poor adherence. Botulinum toxin injection into the bladder wall is invasive, requires re-treatment on a regular basis and carries a risk of urinary retention. Current neuromodulatory techniques are invasive and require highly-specialized care. Therefore, a need exists for a non-invasive, well-tolerated and easily administered therapy for OAB. Transcutaneous spinal cord stimulation (TSCS) has been developed and tested in able bodied individuals to initiate locomotor function as well as in the SCI population for lower extremity and upper extremity function. More recently, we have tested this SCI patients to enable lower urinary tract function and decrease detrusor overactivity, resulting in improved continence.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years
2. Known diagnosis of overactive bladder, confirmed by:

   * presence of urinary frequency, urgency
   * frequent small-volume voids on frequency-volume chart
   * high score on ICIQ-OAB, ICIQ-OABQOL, and OAB-q questionnaires

Exclusion Criteria:

1. Younger than 18 years of age
2. Older than 80 years of age
3. Presence of lower urinary tract symptoms suggestive of urinary retention or obstruction
4. Finding of an elevated post-void residual (>100 ml) on an ultrasonographic bladder scan
5. History of spinal cord injury, spina bifida or other neurological disease affecting the spinal cord
6. Acute or current urinary tract infection
7. History of neuromodulation for overactive bladder (sacral nerve stimulation or peripheral tibial nerve stimulation)
8. Current or planned pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-24 (Estimated); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Number of urination and incontinence episodes over 72 hours | 4-12 weeks
  A voiding diary records the amount of fluid intake, the number of urinations and the number of incontinence episodes over 72 hours. The number of daily urinations and incontinence episodes will be compared at the beginning and the conclusion of the study. Changes in the number of daily urinations and incontinence episodes will be compared between participants in the stimulation and sham arms of the study.
Score on overactive bladder questionnaires | 4-12 weeks
  Each participant will complete two validated questionnaires pertaining to overactive bladder: OAB-q and ICIQ-OAB. The OAB-q generates a total score ranging between 33 points (best) to 198 points (worst). The ICIQ-OAB generates a total score ranging between 0 points (best) to 58 points (worst). The questionnaires will be completed at the initiation and completion of the study. Change in questionnaire scores between initiation and completion of the study will be assessed. Changes in questionnaire scores will be compared between participants in the stimulation and sham arms of the study.

SECONDARY OUTCOMES:
Cystometric bladder capacity, number of detrusor overactivity episodes during urodynamic studies. | 4-12 weeks
  Urodynamic studies will be performed at the initiation and completion of the study. Urodynamic studies will be performed according to ICS (International Continence Society) criteria. Changes in cystometric capacity and number of detrusor overactivity episodes between initiation and completion of the study will be assessed. Changes in these parameters will be compared between participants in the stimulation and sham arms of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Evgeniy I Kreydin, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Background] Irwin DE, Milsom I, Hunskaar S, Reilly K, Kopp Z, Herschorn S, Coyne K, Kelleher C, Hampel C, Artibani W, Abrams P. Population-based survey of urinary incontinence, overactive bladder, and other lower urinary tract symptoms in five countries: results of the EPIC study. Eur Urol. 2006 Dec;50(6):1306-14; discussion 1314-5. doi: 10.1016/j.eururo.2006.09.019. Epub 2006 Oct 2. PMID 17049716
- [Background] Gerasimenko Y, Gorodnichev R, Moshonkina T, Sayenko D, Gad P, Reggie Edgerton V. Transcutaneous electrical spinal-cord stimulation in humans. Ann Phys Rehabil Med. 2015 Sep;58(4):225-231. doi: 10.1016/j.rehab.2015.05.003. Epub 2015 Jul 20. PMID 26205686
- [Background] Gad PN, Kreydin E, Zhong H, Latack K, Edgerton VR. Non-invasive Neuromodulation of Spinal Cord Restores Lower Urinary Tract Function After Paralysis. Front Neurosci. 2018 Jun 29;12:432. doi: 10.3389/fnins.2018.00432. eCollection 2018. PMID 30008661
- [Background] Yoshimura N, Miyazato M, Kitta T, Yoshikawa S. Central nervous targets for the treatment of bladder dysfunction. Neurourol Urodyn. 2014 Jan;33(1):59-66. doi: 10.1002/nau.22455. Epub 2013 Jul 5. PMID 23832777
- [Derived] Zhong H, Liu E, Kohli P, Perez L, Edgerton VR, Ginsberg D, Gad P, Kreydin E. Noninvasive spinal neuromodulation mitigates symptoms of idiopathic overactive bladder. Bioelectron Med. 2022 Mar 23;8(1):5. doi: 10.1186/s42234-022-00087-x. PMID 35317851